CLINICAL TRIAL: NCT04781543
Title: A Randomized, Double-blind, Placebo-controlled, Repeat-dose, Multicenter Trial to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of HZN-825 in Patients With Diffuse Cutaneous Systemic Sclerosis
Brief Title: A Multicenter Trial to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of HZN-825 in Patients With Diffuse Cutaneous Systemic Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to meeting pre-defined criteria for futility.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HZNP-HZN-825-301; 2020-005764-62 (EudraCT Number)
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis; Sclerosis, Systemic
Keywords: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HZN-825 300 mg once daily (QD) (Experimental): One set of 2 HZN-825 150mg tablets in the morning and one set of 2 placebo tablets in the evening.
  Interventions: Drug: HZN-825 QD
- HZN-825 300 mg twice daily (BID) (Experimental): One set of 2 HZN-825 150mg tablets in the morning and one set of 2 HZN-825 150mg tablets in the evening.
  Interventions: Drug: HZN-825 BID
- Placebo (Placebo Comparator): One set of 2 placebo tablets in the morning and one set of 2 placebo tablets in the evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HZN-825 BID — 300 mg oral tablets BID
  Arms: HZN-825 300 mg twice daily (BID)
Drug: Placebo — Placebo BID
  Arms: Placebo
Drug: HZN-825 QD — 300 mg oral tablets QD
  Arms: HZN-825 300 mg once daily (QD)

SUMMARY:
This is a randomized, double-blind, placebo-controlled, repeat-dose, multicenter trial. Participants will be screened within 6 weeks prior to the Baseline (Day 1) Visit. Approximately 300 participants who meet the trial eligibility criteria will be randomized on Day 1 in a 1:1:1 ratio to receive HZN-825 300 mg QD, HZN-825 300 mg BID or placebo for 52 weeks.

The trial will include up to a 42-day Screening Period and a 52-week Double-blind Treatment Period. Participants will take their first dose of trial drug at the clinic and will participate in trial visits at Week 4 and every 6 weeks thereafter until Week 52.

All participants who complete the Double-blind Treatment Period (Week 52) will be eligible to enter a 52-week extension trial (HZNP-HZN-825-302, NCT05626751). Participants not entering the extension trial will participate in a Safety Follow-up Visit 4 weeks after the last dose of trial drug.

DETAILED DESCRIPTION:
Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female between the ages of 18 and 75 years, inclusive, at Screening.
3. Meets the 2013 American College of Rheumatology/European League Against Rheumatism classification criteria for SSc with a total score of ≥9 (Van den Hoogen et al., 2013).
4. Classified as having skin involvement proximal to the elbow and knee (diffuse cutaneous SSc subset by LeRoy and Medsger, 2001).
5. At the time of enrollment, less than or equal to 72 months (6 years) since the onset of the first SSc manifestation, other than Raynaud's phenomenon.
6. Skin thickening from SSc in the forearm suitable for repeat biopsy.
7. mRSS units ≥15 at Screening.
8. FVC ≥45% predicted at Screening, as determined by spirometry.
9. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.

Exclusion Criteria:

1. Positive for anti-centromere antibodies with the exception that subjects who are positive for both anti-centromere and anti-topoisomerase 1 antibodies may be enrolled.
2. Diagnosed with sine scleroderma or limited cutaneous SSc.
3. Diagnosed with other autoimmune connective tissue diseases, except for fibromyalgia, scleroderma-associated myopathy and secondary Sjogren's syndrome.
4. Scleroderma renal crisis diagnosed within 6 months of the Screening Visit.
5. Any of the following cardiovascular diseases:

   1. uncontrolled, severe hypertension (≥160/100 mmHg) or persistent low blood pressure (systolic blood pressure <90 mmHg) within 6 months of Screening,
   2. myocardial infarction within 6 months of Screening,
   3. unstable cardiac angina within 6 months of Screening.
6. DLCO <40% predicted (corrected for hemoglobin). If severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) exposure is of clinical concern for any subject, consider using a DLCO up to 6 months before the Screening Visit.
7. Pulmonary arterial hypertension (PAH) by right heart catheterization requiring treatment with more than 1 oral PAH-approved therapy or any parenteral therapy. Treatment is allowed for erectile dysfunction and/or Raynaud's phenomenon/digital ulcers.
8. Corticosteroid use for conditions other than SSc within 4 weeks prior to Screening (topical steroids for dermatological conditions and inhaled/intranasal/intra-articular steroids are allowed).
9. Use of any other non-steroid immunosuppressive agent, small biologic molecule, cytotoxic or anti-fibrotic drug within 4 weeks of Screening, including cyclophosphamide, azathioprine (Imuran®) or other immunosuppressive or cytotoxic medication. Exceptions include mycophenolate mofetil (CellCept®), mycophenolic acid (Myfortic®), methotrexate and low-dose prednisone, as follows: use of CellCept ≤3 g/day, Myfortic ≤2.14 g/day, methotrexate ≤20 mg/week and prednisone ≤10 mg/day (or equivalent dosing of glucocorticoids) is allowed. Subjects taking CellCept, Myfortic or methotrexate must have been doing so for ≥6 months and the dose must have been stable for ≥4 weeks prior to the Day 1 Visit. Prednisone must have been at a stable dose for ≥8 weeks prior to the Day 1 Visit. It is acceptable to be on background low-dose prednisone and anti-malarial drug along with CellCept, Myfortic or methotrexate. Rituximab must not have been used within 6 months of the Day 1 Visit.
10. Known active bacterial, viral, fungal, mycobacterial or other infection, including tuberculosis or atypical mycobacterial disease (fungal infections of nail beds are allowed) at the time of randomization.
11. Use of a United States Food and Drug Administration-approved agent for SSc or an investigational agent for any condition within 90 days or 5 half-lives, whichever is longer, prior to Screening or anticipated use during the course of the trial.
12. Malignant condition in the past 5 years (except successfully treated basal/squamous cell carcinoma of the skin or cervical cancer in situ).
13. Women of childbearing potential or male subjects not agreeing to use highly effective method(s) of birth control throughout the trial and for 1 month after last dose of trial drug. Male subjects must refrain from sperm donation and females from egg/ova donation for this same time period.
14. Pregnant or lactating women.
15. Current drug or alcohol abuse or history of either within the previous 2 years, in the opinion of the Investigator or as reported by the subject.
16. Previous enrollment in this trial or participation in a prior HZN-825 or SAR100842 clinical trial.
17. Known history of positive test for human immunodeficiency virus (HIV). HIV testing is optional based on Investigator assessment, institutional practices or local guidelines to rule out suspected HIV or potential for a positive HIV result. Subject consent is required prior to HIV testing.
18. Active hepatitis (hepatitis B: positive hepatitis B surface antigen and positive anti-hepatitis B core antibody [anti-HBcAb] and negative hepatitis B surface antibody [HBsAb] or positive for HBcAb with a positive test for HBsAb and with presence of hepatitis B virus DNA at Screening; hepatitis C: positive anti-hepatitis C virus [anti-HCV] and positive RNA HCV).
19. Current alcoholic liver disease, primary biliary cirrhosis or primary sclerosing cholangitis.
20. Previous organ transplant (including allogeneic and autologous marrow transplant).
21. International normalized ratio >2, prolonged prothrombin time >1.5 × the upper limit of normal (ULN) or partial thromboplastin time >1.5 × ULN at Screening.
22. Alanine aminotransferase or aspartate aminotransferase >2 × ULN.
23. Estimated glomerular filtration rate <30 mL/min/1.73 m^2 at Screening.
24. Total bilirubin >2 × ULN. Subjects with documented diagnosis of Gilbert's syndrome may be enrolled if their total bilirubin is ≤3.0 mg/dL.
25. Any other condition that, in the opinion of the Investigator, would preclude enrollment in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Change in FVC (forced vital capacity) percent predicted from Baseline to Week 52 | Baseline to Week 52
  As measured by a pulmonary function test called a spirometry.

SECONDARY OUTCOMES:
Change from Baseline in HAQ-DI (Health Assessment Questionnaire - Disability Index) at Week 52 | Baseline to Week 52
Change from Baseline in MDGA (Physician Global Assessment) at Week 52 | Baseline to Week 52
Change from Baseline in PTGA (Patient Global Assessment) at Week 52 | Baseline to Week 52
Change from Baseline in the Physical Effects subscale of the scleroderma skin patient-reported outcome (SSPRO-18) at Week 52 | Baseline to Week 52
Change from Baseline in the Physical Limitations subscale of the scleroderma skin patient-reported outcome SSPRO-18 at Week 52 | Baseline to Week 52
Proportion of participants with an mRSS (modified Rodnan skin score) decrease of ≥5 points and 25% from Baseline at Week 52 | Baseline to Week 52
Responder rate (defined as ACR-CRISS [predicted probability] of at least 0.6) at Week 52 | Week 52
  American College of Rheumatology-Composite Response Index in Systemic Sclerosis
Proportion of participants with an improvement in ≥3 of 5 core measures from Baseline: ≥20% in mRSS, ≥20% in HAQ-DI, ≥20% in PTGA, ≥20% in MDGA and ≥5% for FVC % predicted at Week 52 (ACR-CRISS-20) | Baseline to Week 52
  American College of Rheumatology-Composite Response Index in Systemic Sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- Serbia (3):
  - Institute of Rheumatology - PPDS, Belgrade
  - Military Medical Academy, Belgrade
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
- Hospital de La Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com